CLINICAL TRIAL: NCT07398365
Title: Medical Phenotyping of NHS General Adult Psychiatry (GAP) Inpatients
Status: Recruiting | Type: Observational
Sponsor: University of Edinburgh (Other)
Collaborators: University of Dundee (Other); NHS Lothian (Other Government)
Responsible Party: Sponsor
Other Study IDs: 337967
Record Dates: First submitted 2025-09-24; First posted 2026-02-09 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2025-09

CONDITIONS: Bipolar Affective Disorder; Schizophrenia Disorders; Depression Disorders; Personality Disorders
Keywords: General Adult Psychiatry; mental health; physical health; inpatients; schizophrenia; NHS; Bipolar affective disorder; depression; psychosis; treatment resistance; personality disorder; cardiometabolic disease; cancer; respiratory disease
MeSH Terms: conditions — Bipolar Disorder; Schizophrenia; Personality Disorders; Psychological Well-Being; Depression; Psychotic Disorders; Neoplasms; Respiration Disorders | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Group 1 - Schizophrenia Group: * Schizophrenia - 6A20
  * Schizoaffective disorder - 6A21
  * Delusional disorder - 6A24
  * Other primary psychotic disorders (psychosis NOS) - 6A2Z
  * Schizotypal disorder - 6A23
  Interventions: Other: Questionnaires, rating scales, & review of notes
- Group 2 - Bipolar Group: * Bipolar type I disorder, current episode manic - 6A60 • without psychotic symptoms - 6A60.0 • with psychotic symptoms - 6A60.2
  * Bipolar type II disorder, current episode depressed, with psychotic symptoms - 6A60.6
  Interventions: Other: Questionnaires, rating scales, & review of notes
- Group 3 -Depression Group: * Recurrent depressive disorder, current severe episode without psychotic symptoms - 6A71.3
  * Single episode depressive disorder, moderate with psychotic symptoms - 6A70.2
  * Recurrent depressive disorder (not otherwise specified) - 6A71
  * Mixed depressive and anxiety disorder - 6A73
  Interventions: Other: Questionnaires, rating scales, & review of notes
- Group 4 - Personality Group: * Personality disorder - 6D10, 6D10.Z
  * Complex post-traumatic stress disorder - 6B41
  * Substance use disorders - 6C4* codes (e.g., 6C4G.1 alcohol, 6C45.6 sedative-hypnotic, 6C43.2 cannabis, 6C44.2 stimulants, 6C4Z unspecified)
  Interventions: Other: Questionnaires, rating scales, & review of notes

INTERVENTIONS:
Other: Questionnaires, rating scales, & review of notes — Observational - questionnaires, rating scales, & review of notes

SUMMARY:
This observational study will characterise the general psychiatric and general medical phenotypes of 100 adults, sequentially admitted to NHS General Adult Psychiatry (GAP) "mental health" inpatient wards, providing the first detailed information on morbidity in this patient population.

DETAILED DESCRIPTION:
It is often supposed that most patients who attend secondary care General Adult Psychiatry (GAP) services would be excluded from clinical trials because they have too many co-morbidities, they are 'treatment resistant' (have a condition that does not improve despite trying two or more standard treatments), and their conditions are too severe. Hence, it would be helpful to properly measure these variables in GAP patients using questionnaires and a review of the case notes to see how many GAP patients would indeed be excluded from clinical trials. It is anticipated that this will show that the participants in clinical trials are very different from 'real life' GAP patients, and that could explain why some promising results from clinical trials do not translate into useful new treatments. Also, this data could act as a benchmark or baseline against which to measure the efficacy of novel treatments and interventions.

PRIMARY OBJECTIVE

Using the most commonly employed diagnostic tools, severity rating scales, and a systematic review of the case notes, the typical characteristics of GAP patients will be described.

SECONDARY OBJECTIVES

The above data will be used to compared 'typical/real life' patients with the participants in impactful clinical trials.

This is a cross sectional quantitative study. Participants will spend about an hour attending to the questionnaires and talking to their clinician.

STUDY SETTING

The study will take place in St John's Hospital, Livingston, West Lothian, on the acute psychiatric ward, and the outpatient department.

STUDY POPULATION

100 patients who attend the West Lothian NHS GAP service will be consecutively recruited. These participants will be between 18 and 65 years old and suffering from mental disorders that their GP could not treat.

IDENTIFYING PARTICIPANTS

The usual clinical team will ask eligible patients if they would like to participate.

CONSENTING PARTICIPANTS

Consent will be thoroughly informed by an information leaflet and subsequent discussion with the involved clinician. Participants will take the information leaflet away with them and express their consent, or not, in their own time by using the contact details on the information leaflet, or when they next see their clinician.

WITHDRAWAL OF STUDY PARTICIPANTS

Participants will have the option of withdrawal from all aspects of the trial, but the data collected up to that point could be used. To safeguard rights, the minimum personally identifiable information possible will be collected. There are no stopping rules. Participants could withdraw at any time.

ELIGIBILITY:
Inclusion:

- Adults aged between 18 and 65 years admitted to GAP wards during recruitment period

Exclusion:

- Admissions to non-GAP wards (e.g., forensic psychiatry, young people's units, perinatal, old age psychiatry, or general medical wards)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults (≥18 years) consecutively admitted to NHS GAP inpatient wards in Scotland.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2024-04-03 (Actual); Primary Completion 2026-04-03 (Estimated); Study Completion 2026-08-08 (Estimated)

PRIMARY OUTCOMES:
Rates of comorbid physical illnesses | At enrolment
  As per medical note review and physical examination - BMI
Psychiatric diagnosis | At enrolment
  ICD-11 codes
Severity of psychosis | At enrolment
  Brief Psychiatric Rating Scale (BPRS) score; 18 to 126, higher scores indicate more severe symptoms
Depression of severity | At enrolment
  Inventory of Depressive Symptomatology Self Report (IDS-SR); 0 to 84, higher scores indicate more severe symptoms
Severity of mania | At enrolment
  Young Mania Rating Scale score; 0 to 60, higher scores indicate more severe symptoms
Severity of anxiety | At enrolment
  General Anxiety Scale (GAD-7) score; 0 to 21, higher scores indicate more severe symptoms
Substance use | At enrolment
  Tobacco, Alcohol, Prescription medication, and other Substance use (TAPS) tool score; tobacco 0 to 3, alcohol 0 to 4, others 0 to 21, higher scores indicate more risky use
Mental Health Act status | At enrolment
  MHA detention status; informal or detained
Treatment resistance indicators | At enrolment
  Clozapine for psychosis, and ECT treatment and Massachusetts General Hospital Staging (MGH-S) score for depression. MGH-S uses the number of failed trials with the intensity/optimization of each trial to produce a score where >3.5 defines treatment resistant depression
Rates of abnormal findings on physical examination | At enrolment
  When psychiatric patients are admitted to hospital, they are examined by a resident doctor, including inspection, auscultation, and palpation. Rates of abnormal findings on cardiovascular , respiratory, abdominal, and neurological examination will be noted..
Abnormal laboratory values | At enrolment
  When psychiatric patients are admitted to hospital, screening blood tests, including full blood count, urea and electrolytes (kidney), liver function tests, random glucose, cholesterol, triglycerides, and thyroid function tests.
Rates of comorbid physical illness | At enrolment
  As per medical note review and physical examination - blood pressure mmHg
Rates of comorbid physical illness | At enrolment
  As per medical note review and physical examination - cardiometabolic disease
Rates of comorbid physical illness | At enrolment
  As per medical note review and physical examination - neurological disease.
Rates of comorbid physical illness | At enrolment
  As per medical note review and physical examination - musculoskeletal disease
Rates of comorbid physical illness | At enrolment
  As per medical note review and physical examination - respiratory disease
Rates of comorbid physical illness | At enrolment
  As per medical note review and physical examination - renal disease
Rates of comorbid physical illness | At enrolment
  As per medical note review and physical examination - hepatic disease
Rates of comorbid physical illness | At enrolment
  As per medical note review and physical examination - haematological disease

CONTACTS AND LOCATIONS:
Overall Officials: Douglas Steele, Study Director — University of Dundee
Locations (1):
- St John's Hospital, Livingston, West Lothian, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Anonymous data only - diagnosis (ICD-11 codes), severity ratings (BPRS, IDS-SR, YMRS, Hamilton scales), MHA detention status, treatment resistance indicators (e.g., clozapine, ECT treatment, MGH-S), comorbid physical diagnoses, abnormal findings on physical examination, abnormal laboratory values, cardiometabolic measures
Access Criteria: Anonymous data available to co-investigators - diagnosis (ICD-11 codes), severity ratings (BPRS, IDS-SR, YMRS, Hamilton scales), MHA detention status, treatment resistance indicators (e.g., clozapine, ECT treatment, MGH-S), comorbid physical diagnoses, abnormal findings on physical examination, abnormal laboratory values, cardiometabolic measures